CLINICAL TRIAL: NCT06506240
Title: Effects of Acupuncture for Senile Pruritus: Study Protocol for a Randomised Controlled Trial
Brief Title: Effects of Acupuncture for Senile Pruritus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, He Chen, Mr., Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-087-KY
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Senile Pruritus
Keywords: Acupuncture; Senile pruritus; Randomized controlled trial
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This trial is a single-center, parallel-arm, randomized, sham-controlled clinical trial. Eligible participants are randomized and allocated to either the acupuncture or sham acupuncture groups at a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients meeting the eligibility criteria for SP will be randomly assigned to either the acupuncture or sham acupuncture groups in a 1:1 ratio. The randomization sequence was generated using the blockrand package in R software (version 4.1.1) and is detailed in the supplementary materials. The sequence will be enclosed in sealed, opaque, sequentially numbered envelopes, which will be opened after participants complete all baseline assessments. Allocation to the assigned group will be conducted by a research assistant who is not involved in treatment or outcome assessments. Participants, outcome assessors, and the statistician will be blinded to group assignments, ensuring unbiased evaluation. However, the practitioner administering the intervention will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Experimental): Treatment will be administered by licensed practitioners with over five years of experience, in separate rooms to prevent patient interaction. The selected acupuncture points include LI11 , SP10, ST36, SP6, LR3, LI4, ST25, CV4, GV20, and superior GV29. Sterile disposable stainless-steel needles (0.3 mm×40 mm; Hwato brand, Suzhou Medical Appliance Factory, Suzhou, China) will be used. Patients will lie supine, and routine skin sterilization will be performed locally. Needles will be inserted at depths ranging from 10 to 30 mm at the designated acupuncture points. Each needle will be manually manipulated with lifting, thrusting, twirling, and rotating to elicit Deqi sensation (including soreness, numbness, distention, and heaviness). Needles will remain inserted for 30 minutes per session and manipulated three times, every 10 minutes. Acupuncture sessions will be conducted three times weekly over a six-week period.
  Interventions: Other: Acupuncture
- Sham acupuncture group (Sham Comparator): Patients in the control group will undergo sham acupuncture using sterile disposable stainless-steel needles (0.3 mm×25 mm; Hwato brand, Suzhou Medical Appliance Factory, Suzhou, China). Needles will be inserted to depths of 2 to 3 mm at the same acupuncture points as in the acupuncture group. There will be no needle manipulation or attempt to induce Deqi sensation. Needles will be retained for 30 minutes per session.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Treatment will be administered by licensed practitioners with over five years of experience, in separate rooms to prevent patient interaction. The selected acupuncture points include LI11 (Quchi), SP10 (Xuehai), ST36 (Zusanli), SP6 (Sanyinjiao), LR3 (Taichong), LI4 (Hegu), ST25 (Tianshu), CV4 (Guanyuan), GV20 (Baihui), and superior GV29 (superior Yintang). Patients will receive acupuncture or sham acupuncture three times weekly for 6 weeks.

SUMMARY:
Senile pruritus (SP), characterized by idiopathic itching in individuals aged 60 years and older without primary skin lesions, significantly impacts sleep and quality of life. Effective alternative treatments are needed. Acupuncture has been suggested as a potential intervention to alleviate itching; however, its role in managing SP remains uncertain. This study aims to evaluate the effects and safety of acupuncture for SP. This single-centre, parallel, two-arm, randomized, sham-controlled trial will enroll 108 patients diagnosed with SP in a 1:1 ratio to either the acupuncture or sham acupuncture group. Participants, outcome assessors, and the statistician will be blinded. Treatment will consist of 18 sessions over 6 weeks. The primary outcome is change from baseline in the Numerical Rating Scale (NRS) score for average itching severity at week 6, assessed weekly via weekly diary of pruritus assessment. Secondary outcomes include changes in NRS score for maximum itching severity, daily episodes of itching, itchy area of body surface, overall dry skin score (ODS), the Dermatology Life Quality Index (DLQI), the Pittsburgh Sleep Quality Index (PSQI), the Hospital Anxiety and Depression Scale (HADS), and Patient Global Impression of Change (PGIC). Adverse events will be monitored throughout the study period. The intention-to-treat (ITT) population will include participants who complete baseline assessments and receive at least one treatment session.

ELIGIBILITY:
Inclusion Criteria:

Participants aged between 60 and 80 years who meet diagnostic criteria for SP, with an average severity score of itching in the past week of ≥4 points on the Numerical Rating Scale (NRS), and who voluntarily provide written informed consent are eligible for inclusion.

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

1. Severe skin damage or infection;
2. Severe underlying diseases including cardiovascular diseases, hepatobiliary diseases, kidney diseases, hematologic diseases, autoimmune diseases, infectious diseases, severe malnutrition, or malignancies;
3. Mental illness, cognitive dysfunction, or language disorders;
4. Received acupuncture therapy for pruritus within the past month;
5. Have a history of drug abuse.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Numeric Rating Scale (NRS) scores for average itching severity at week 6. | Week 6
  This will be assessed using weekly diaries for pruritus evaluation.

SECONDARY OUTCOMES:
Change from baseline in NRS score for average itching severity | Week 2, 4, 10, 14, and 18
  Assessed through weekly diary of pruritus assessment
Change from baseline in NRS score for maximum itching severity | Week 2, 4, 6, and week 10, 14, and 18
  Assessed through weekly diary of pruritus assessment
Number of episodes of itching per day | Week 2, 4, 6, and week 10, 14, and 18
  Assessed through weekly diary of pruritus assessment
Change from baseline in itchy area of the body surface | Week 6, 10, 14, and 18
  Measured using the Chinese Rule of Nine
ODS | Week 6, 10, 14, and 18
  ODS
Change from baseline in DLQI | Week 6, 10, 14, and 18
  Change from baseline in DLQI
Change from baseline in PSQI | Week 6, and 18
  Change from baseline in PSQI
Change from baseline in HADS | Week 6, and 18
  Change from baseline in HADS
PGIC | Week 6, and 18
  PGIC

OTHER OUTCOMES:
Adverse events | Week 0 to week 18
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, informed consent form (ICF) will be shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Chen H, Liu S, Gao S, Yi J, Shi H, Fang J, Wang W, Chen H, Liu Z. Effects and safety of acupuncture versus non-penetrating sham acupuncture for senile pruritus: Rationale and design for a randomized controlled trial. Contemp Clin Trials Commun. 2025 Feb 12;44:101454. doi: 10.1016/j.conctc.2025.101454. eCollection 2025 Apr. PMID 40027278